CLINICAL TRIAL: NCT06291376
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Ravulizumab in Adult Participants With Immunoglobulin A Nephropathy (IgAN)
Brief Title: Study of Ravulizumab in Immunoglobulin A Nephropathy (IgAN)
Acronym: ICAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D928FC00001
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Immunoglobulin A Nephropathy; IgAN
Keywords: Immunoglobulin A nephropathy; IgAN; proteinuria; glomerulonephropathy; chronic kidney disease; CKD
MeSH Terms: conditions — Glomerulonephritis, IGA; Proteinuria; Renal Insufficiency, Chronic | interventions — ravulizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ravulizumab IV q8w (Experimental): Participants will receive a weight-based loading dose on Day 1 followed by weight-based maintenance dosing initiated on Day 15, and then administered every 8 weeks (q8w).
  Interventions: Drug: Ravulizumab
- Placebo IV q8w (Placebo Comparator): Participants will receive a weight-based loading dose on Day 1 followed by weight-based maintenance dosing initiated on Day 15, and then administered q8w.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ravulizumab — Participants will receive ravulizumab via weight-based intravenous (IV) infusion.
  Arms: Ravulizumab IV q8w
Drug: Placebo — Participants will receive placebo via weight-based IV infusion.
  Arms: Placebo IV q8w

SUMMARY:
The primary objective of this study to evaluate efficacy of ravulizumab compared with placebo on proteinuria reduction and change in eGFR in adult participants with IgAN who are at risk of disease progression.

DETAILED DESCRIPTION:
The I CAN study will enroll approximately 510 eligible participants with IgAN who are high risk of disease progression. Participants will be on stable concomitant IgAN treatment(s) consistent with standard of care for patients with IgAN for at least 3 months prior to Screening. Approximately 450 participants will be randomized in a 1:1 allocation ratio to receive a weight-based IV infusion of either ravulizumab or placebo. An interim analysis may be conducted at Week 34 to evaluate change in proteinuria and the final analysis will be conducted at Week 106 to evaluate eGFR. In addition, approximately 60 participants with eGFR 20-29 mL/min/1.73m2 will be enrolled in an Advanced Kidney Disease (AdKD) Cohort After Week 106, all participants have the option to enter an Open-label Ravulizumab Access Period.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of IgAN diagnosis established on kidney biopsy obtained any time prior to or during the Screening Period for participants with eGFR ≥ 30 mL/min/1.73 m^2.
* For participants in the AdKD cohorts, eGFR 20 to 29 mL/min/1.73 m2 a kidney biopsy is required within 6 months prior to Screening or during the Screening Period.
* UPCR ≥ 0.75 g/g or UP ≥1 g/day calculated from the mean of two 24-hour urine during the Screening Period.
* Estimated GFR ≥ 30 mL/min/1.73 m2 at Screening.
* Stable and maximum allowed or tolerated RASI (ACEI and/or ARB) dose for ≥ 3 months prior to Screening with no planned change during Screening through Week 106.
* Participants who are receiving SGLT2I, DEARA, MRA or ERA must be on a stable and maximum allowed or tolerated dose for ≥ 3 months prior to Screening with no planned change in dose through Week 106.

Exclusion Criteria:

* Diagnosis of rapid progressive glomerulonephritis as measured by eGFR loss ≥ 50% over a period of 3 months prior to Screening.
* Secondary IgAN (eg, due to systemic lupus erythematosus (SLE), cirrhosis, or celiac disease; IgAV-N may be eligible).
* Concomitant clinically significant renal disease other than IgAN.
* Prior use of immunosuppressive treatment within 3 months of screening.
* Uncontrolled diabetes mellitus with glycosylated hemoglobin (HbA1c) > 8.5%.
* Henoch-Schonlein purpura (IgAV) requiring systemic immunosuppressive therapy within 12 months of Screening.
* History of kidney transplant or planned kidney transplant during the Treatment Period.
* Splenectomy or functional asplenia.
* History of Neisseria meningitidis infection.
* Active systemic bacterial, viral, or fungal infection within 14 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2030-07-19 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Proteinuria Based on 24-hour Urine Protein Creatinine Ratio (UPCR) at Week 34 | Baseline, Week 34
  Evaluated at interim analysis only
Change from Baseline in Glomerular Filtration Rate (eGFR) at Week 106 | Baseline, Week 106
  Evaluated at final analysis only

SECONDARY OUTCOMES:
Change from Baseline in Proteinuria Based on 24-hour Urine Protein Creatinine Ratio (UPCR) at Weeks 10, 26, 34, 50, and 106 | Baseline, Weeks 10, 26, 34, 50, and 106
  Evaluated at interim and final analysis
Change From Baseline in eGFR at Weeks 34 and 50 | Baseline, Weeks 34 and 50
  Evaluated at interim and final analysis
Change From Baseline in Albuminuria at Each Scheduled Visit Up to Week 106 | Baseline, at Each Scheduled Visit Up to Week 106
  Evaluated at interim and final analysis
Reduction in 24-hour UPCR ≥ 50% From Baseline at Each Scheduled Visit Up to Week 106 | Baseline, at Each Scheduled Visit Up to Week 106
  Evaluated at interim and final analysis
Number of Participants With Partial Remission at Each Scheduled Visit Up to Week 106 | Baseline, at Each Scheduled Visit Up to Week 106
  Evaluated at interim and final analysis
Change from Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue at Weeks 34, 50, and 106 | Baseline, Weeks 34, 50, and 106
  Evaluated at interim and final analysis
Annualized eGFR Slope Over 50 Weeks | Baseline, Over 50 Weeks
  Evaluated at interim analysis only
Time to First Composite Kidney Event Up to Week 106 | Baseline Up to Week 106
  Composite kidney event endpoint is defined as reaching at least 1 of the following: Sustained ≥ 30% decline in eGFR relative to baseline; or Sustained eGFR < 15 milliliter (mL)/minute (min)/1.73 square meter (m^2); or Maintenance dialysis; or Receipt of kidney transplant; or Death from kidney failure.
  Evaluated at final analysis only
Time to Sustained ≥ 30% eGFR Decline Up to Week 106 | Baseline Up to Week 106
  Evaluated at final analysis only
Time to Sustained eGFR Decline ≥ 40% Up to Week 106 | Baseline Up to Week 106
  Evaluated at final analysis only
Use of Alternative IgAN Therapy Up to Week 106 | Baseline, Up to Week 106
  Evaluated at final analysis only

CONTACTS AND LOCATIONS:
Locations (271):
- United States (43):
  - Research Site, Alabaster, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Bernardino, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Stanford, California
  - Research Site, Torrance, California
  - Research Site, Valencia, California
  - Research Site, Aurora, Colorado
  - Research Site, Bay Pines, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Acworth, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Iowa City, Iowa
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Augusta, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Pontiac, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, City of Saint Peters, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, North Las Vegas, Nevada
  - Research Site, Albany, New York
  - Research Site, East Setauket, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Columbus, Ohio
  - Research Site, Charleston, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Shenandoah, Texas
  - Research Site, Temple, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Milwaukee, Wisconsin
- Argentina (6):
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Rosario
  - Research Site, San Juan Bautista
  - Research Site, San Luis
- Australia (10):
  - Research Site, Camperdown
  - Research Site, Canberra
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, Herston
  - Research Site, Liverpool
  - Research Site, Parkville
  - Research Site, Perth
  - Research Site, Southport
  - Research Site, St Albans
- Austria (3):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Linz
- Belgium (5):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
- Brazil (9):
  - Research Site, Belo Horizonte
  - Research Site, Botucatu
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Recife
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (5):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Brampton, Ontario
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- Chile (4):
  - Research Site, Araucania
  - Research Site, Providencia
  - Research Site, Santiago
  - Research Site, Valdivia
- China (29):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changzhou
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Lanzhou
  - Research Site, Luoyang
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Yantai
  - Research Site, Yibin
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
  - Research Site, Zhongshan
- Colombia (6):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Manizales
  - Research Site, Medellín
  - Research Site, Rionegro
- Czechia (2):
  - Research Site, Nový Jičín
  - Research Site, Prague
- France (13):
  - Research Site, Amiens
  - Research Site, Bayonne
  - Research Site, Brest
  - Research Site, Chambéry
  - Research Site, Clermont-Ferrand
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Nice
  - Research Site, Paris
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (11):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Greifswald
  - Research Site, Hanover
  - Research Site, Konstanz
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Villingen-Schwenningen
- Greece (4):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Lai Chi Kok
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Miskolc
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Nazareth
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
- Italy (13):
  - Research Site, Agrigento
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Cagliari
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Piacenza
  - Research Site, Torino
  - Research Site, Torrette
  - Research Site, Verona
- Japan (15):
  - Research Site, Ashikaga
  - Research Site, Bunkyō City
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Kamakura
  - Research Site, Kasugai-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Kobe
  - Research Site, Matsumoto-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Toyota-Shi
  - Research Site, Urayasu-shi
- Malaysia (5):
  - Research Site, Ipoh
  - Research Site, Johor Bahru
  - Research Site, Kuala Lumpur
  - Research Site, Seremban
  - Research Site, Taiping
- Mexico (6):
  - Research Site, Chihuahua City
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Juriquilla
  - Research Site, México
  - Research Site, Zapopan
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (5):
  - Research Site, Braga
  - Research Site, Funchal
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Torres Novas
- Romania (3):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Timișoara
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Martin
- South Korea (7):
  - Research Site, Anyang-si
  - Research Site, Busan
  - Research Site, Deagu
  - Research Site, Gwangju
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (12):
  - Research Site, A Coruña
  - Research Site, Alcalá de Henares
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Oviedo
  - Research Site, Sant Joan Despí
  - Research Site, Seville
  - Research Site, Tarragona
  - Research Site, Valencia
  - Research Site, Zaragoza
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chaingmai
  - Research Site, Khlong Luang
  - Research Site, Khon Kaen
- Turkey (Türkiye) (8):
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
  - Research Site, Konya
  - Research Site, Pamukkale
- United Kingdom (9):
  - Research Site, Cambridge
  - Research Site, Doncaster
  - Research Site, Dundee
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Reading
  - Research Site, Salford
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Lafayette R, Tumlin J, Fenoglio R, Kaufeld J, Perez Valdivia MA, Wu MS, Susan Huang SH, Alamartine E, Kim SG, Yee M, Kateifides A, Rice K, Garlo K, Barratt J; SANCTUARY Study Investigators. Efficacy and Safety of Ravulizumab in IgA Nephropathy: A Phase 2 Randomized Double-Blind Placebo-Controlled Trial. J Am Soc Nephrol. 2025 Apr 1;36(4):645-656. doi: 10.1681/ASN.0000000534. Epub 2024 Oct 25. PMID 39455063